CLINICAL TRIAL: NCT05116865
Title: A Double-Blinded, Randomized, and Placebo-Controlled Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetics Profile of Single and Multiple Ascending Doses of Inhaled HH-120 Aerosol in Healthy Volunteers
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Inhaled HH-120 Aerosol in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HH120-101
Record Dates: First submitted 2021-10-19; First posted 2021-11-11 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: COVID-19 Respiratory Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Single Ascending Dose Cohort A1 (Experimental): Subjects will receive a single dose of either dose level 1 of HH-120 or placebo
  Interventions: Biological: HH-120 Dose 1; Drug: Placebo
- Single Ascending Dose Cohort A2 (Experimental): Subjects will receive a single dose of either dose level 2 of HH-120 or placebo
  Interventions: Biological: HH-120 Dose 2; Drug: Placebo
- Single Ascending Dose Cohort A3 (Experimental): Subjects will receive a single dose of either dose level 3 of HH-120 or placebo
  Interventions: Biological: HH-120 Dose 3; Drug: Placebo
- Multiple Ascending Doses Cohort B1 (Experimental): Subjects will receive multiple doses of either Dose level 1of HH-120 or placebo
  Interventions: Biological: HH-120 Dose 1; Drug: Placebo
- Multiple Ascending Doses Cohort B2 (Experimental): Subjects will receive multiple doses of either Dose level 2 of HH-120 or placebo
  Interventions: Biological: HH-120 Dose 2; Drug: Placebo
- Multiple Ascending Doses Cohort B3 (Experimental): Subjects will receive multiple doses of either Dose level 3 of HH-120 or placebo
  Interventions: Biological: HH-120 Dose 3; Drug: Placebo

INTERVENTIONS:
Biological: HH-120 Dose 1 — Dose level 1 of HH-120
  Other Names: HH-120
  Arms: Multiple Ascending Doses Cohort B1; Single Ascending Dose Cohort A1
Biological: HH-120 Dose 2 — Dose level 2 of HH-120
  Other Names: HH-120
  Arms: Multiple Ascending Doses Cohort B2; Single Ascending Dose Cohort A2
Biological: HH-120 Dose 3 — Dose level 3 of HH-120
  Other Names: HH-120
  Arms: Multiple Ascending Doses Cohort B3; Single Ascending Dose Cohort A3
Drug: Placebo — Placebo to match

SUMMARY:
This is a Phase 1, randomized, double-blinded, placebo controlled, dose escalation study of HH-120 in healthy adult volunteers. HH-120 is a novel inhalable biologic being developed for COVID-19 treatment. The study aims to evaluate the safety, tolerability and pharmacokinetic profile of HH-120 administered by aerosol inhalation after single and multiple ascending doses.

DETAILED DESCRIPTION:
Approximately 48 participants will be sequentially enrolled into either 1 of 3 SAD cohorts (n=8 per cohort), or 1 of 3 MAD cohorts (n= 8 per cohort). An adaptive dose escalation schedule will be employed for both SAD and MAD parts of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers aged 18 to 65 years (both inclusive)
2. Participants must have a body mass index between ≥ 18.0 and ≤ 32 .0 kg/m2 and a bodyweight of at least 45 kg at Screening.
3. Participants must be a non-smoker and must not have used any tobacco products within 90 days prior to Screening.
4. Participants must be in good general health, with no significant medical history, have no clinically significant abnormalities on physical examination at screening and/or before administration of the initial dose of IP.
5. Participants must have clinical laboratory values within normal range.
6. Females must be non-pregnant and non-lactating, and must use an acceptable, highly effective double contraception from Screening until study completion, including the follow-up period.
7. Males must not donate sperm for at least 90 days after the last dose of IP.
8. Participants must have the ability and willingness to attend the necessary visits to the CRU.

Exclusion Criteria:

1. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period.
2. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the PI's (or delegate's) opinion, could adversely affect the safety of the participant or that might interfere with the conduct of the study.
3. Presence of any underlying physical or psychological medical condition
4. Pre-existing severe obstructive disease of the respiratory system such as chronic obstructive pulmonary disease or asthma , including resolved childhood asthma, which may impact inhalation as judged by the PI, delegate, or Sponsor.
5. History or evidence o f any anatomical airway defect, which in the opinion of the PI, may impact inhalation.
6. Abnormal spirometry findings at Screening that are considered by the PI to be clinically significant, including FEV1 < 80% or FVC < 80%.
7. Blood donation of > 500 mL or significant blood loss within 60 days prior to the first IP administration or plasma donation within 7 days prior to IP administration.
8. Systemic or respiratory infection within 2 weeks before the Screening visit or fever (tympanic temperature > 37.5°C) or symptomatic viral or bacterial infection at time of Screening.
9. Current infection with SARS-CoV-2, infection within the 2 weeks prior to Screening, or a history of SARS-CoV-2 infection plus symptoms of post-COVID syndrome.
10. History of anaphylaxis or other significant allergy in the opinion of the PI or known allergy or hypersensitivity to any of the components of the IP.
11. History of malignancy, except for non-melanoma skin cancer, excised more than 2 years ago and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening.
12. A personal history of unexplained blackouts or fainting or known risk factors for Torsade de Pointes (eg, hypokalemia, heart failure).
13. Abnormal 12-lead ECG findings at Screening that are considered by the PI to be clinically significant, including arrhythmias or marked QT interval abnormalities (QTcF < 300 msec or ≥ 450 msec at Screening).
14. Confirmed (eg, 2 consecutive triplicate measurements) average systolic blood pressure (SBP) > 140 or < 90 mmHg, and diastolic blood pressure (DBP) > 90 or < 45 mmHg at Screening.
15. Confirmed (eg, 2 consecutive triplicate measurements) average resting HR > 100 or < 45 beats per minute at Screening.
16. Vaccination with a live vaccine within the 4 weeks prior to Screening or that is planned within 4 weeks of dosing, and any non-live vaccination within the 2 weeks prior to Screening, or that is planned within 2 weeks of dosing or planned during study participation (including vaccines for COVID-19).
17. Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody at Screening.
18. Participants with a positive toxicology screening panel (urine test including qualitative identification of barbiturates, tetrahydrocannabinol [THC], amphetamines, benzodiazepines, opiates, cocaine, and cotinine), or alcohol breath test at Screening or Day -1.
19. Participants with a history of substance abuse or dependency or history of recreational intravenous (IV) drug use over the last 6 months (by self-declaration).
20. Use of any IP or medical device within 30 days prior to screening.
21. Use of any prescription drugs for 14 days prior to dosing or over the counter medication, herbal remedies, supplements or vitamins 7 days prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) | Day 1- Day 15 (SAD) or Day 22 (MAD)
  An Adverse Event (AE) is any event, side-effect or any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE that started on or after the first study treatment or that worsened after the first study treatment will be regarded as TEAEs.
Severity of treatment emergent adverse events (TEAEs)as assessed by CTCAE v5.0 | Day 1- Day 15 (SAD) or Day 22 (MAD)
  An Adverse Event (AE) is any event, side-effect or any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE that started on or after the first study treatment or that worsened after the first study treatment will be regarded as TEAEs.
Duration of treatment emergent adverse events (TEAEs) | Day 1- Day 15 (SAD) or Day 22 (MAD)
  An Adverse Event (AE) is any event, side-effect or any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE that started on or after the first study treatment or that worsened after the first study treatment will be regarded as TEAEs.
Number of participants with serious adverse events (SAEs) | Day 1- Day 15 (SAD) or Day 22 (MAD)
  A serious adverse event (SAE) is defined as an AE occurring during any study phase and at any dose of IP (active or placebo) that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect
Severity of serious adverse events (SAEs) as assessed by CTCAE v5.0 | Day 1- Day 15 (SAD) or Day 22 (MAD)
  A serious adverse event (SAE) is defined as an AE occurring during any study phase and at any dose of IP (active or placebo) that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect
Duration of serious adverse events (SAEs) | Day 1- Day 15 (SAD) or Day 22 (MAD)
  A serious adverse event (SAE) is defined as an AE occurring during any study phase and at any dose of IP (active or placebo) that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect
Number of participants with abnormal clinically significant physical examination findings | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Complete and symptom directed physical examination will be performed
Number of participants with abnormal clinically significant electrocardiogram (ECG) | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Single resting 12- lead ECGs will be collected
Number of participants with clinically significant change in vital signs from baseline | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Vital signs include heart rate, blood pressure, respiratory rate and tympanic temperature
Changes in the spirometry score from Baseline | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Measured by Forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1) after dosing
Number of participants with abnormal clinically significant clinical laboratory parameters | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Clinical laboratory test include hematology, coagulation, biochemistry and urinalysis

SECONDARY OUTCOMES:
Cmax in SAD and MAD | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Maximum observed HH-120 concentration
Tmax in SAD and MAD | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Time to the maximum observed HH-120 concentration
t1/2 in SAD and MAD part | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Terminal elimination half life calculated as ln (2)/λz
AUC0-last | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Area under the plasma concentration-time curve from time zero (from the start of inhalation time) to the last time point with measurable analyte concentration
AUC0-inf | Day 1- Day 15 (SAD) or Day 22 (MAD)
  AUC from time zero (from the start of inhalation time) extrapolated to infinity
%AUCextrap | Day 1- Day 15 (SAD) or Day 22 (MAD)
  The percentage of the AUC that has been extrapolated beyond the last observed data point
Kel or λz | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Apparent terminal elimination rate constant, calculated by linear regression of the terminal linear portion of the log concentration vs time curve
CL/F | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Apparent total body clearance
Vz/F in SAD | Day 1- Day 15 (SAD) or Day 22 (MAD)
  Apparent volume of distribution during the terminal phase
CL/Fss in MAD | Day 1-Day 22
  Apparent total plasma clearance at steady state
Vz/Fss in MAD | Day1- Day 22
  Apparent terminal volume of distribution at steady state
Accumulation ratio (RA) | Day 1- Day 7
  AUC0-24 hours on Day 7/AUC0-24 hours on Day 1
Immunogenicity of HH-120 | Day 1- Day 15 (SAD) or Day 22 (MAD)
  To determine the presence and levels of anti-drug antibody (ADA).

CONTACTS AND LOCATIONS:
Overall Officials: Yongqing Lin, Study Director — Huahui Health Ltd
Locations (1):
- Nucleus Network, Brisbane, Queensland, Australia